CLINICAL TRIAL: NCT07323771
Title: The Effectiveness of Educational Intervention Based on Health Belief Model Delivered Via WhatsApp on Oral Health Knowledge and Behaviors of Individuals With Type 2 Diabetes Mellitus; A Randomized Controlled Trial
Brief Title: Improving Oral Health Knowledge and Habits in People With Diabetes Through a Theory Guided WhatsApp Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, ILMA KIRAN, MPH Trainee and Lecturer, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB4057/DUHS/Approval/2025/294
Record Dates: First submitted 2025-12-08; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Oral Health Knowledge; Oral Health Behavior Change; Diabetes Type 2
Keywords: Type 2 Diabetes Mellitus; Dental Health Education; Health Belief Model; Digital Health; Social Media
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Health Belief Model

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the intervention group or the control group, following a 1:1 allocation ratio. The randomization process was stratified based on three key characteristics including gender, educational level, and duration of diabetes, to ensure balanced distribution and to minimize potential bias.
  Randomization was conducted using random number generator where each participant was assigned a random number, then participants were allocated equally into either Intervention Group which received HBM based education via WhatsApp or control Group which received an educational brochure.
Who Masked: Participant
Masking Description: This study was single blinded in which participants were not informed about the presence of two distinct groups; they were only aware about receiving education related to oral health.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Brochure Group (Other): Participants in this group receive oral health education through an educational brochure
  Interventions: Behavioral: Educational Brochure Group
- Health Belief Model Based WhatsApp Oral Health Education Program (Other): Participants receive a Health Belief Model (HBM) based oral health education program through WhatsApp videos for four weeks.
  Interventions: Behavioral: Health Belief Model (HBM) Based WhatsApp Oral Health Education Program

INTERVENTIONS:
Behavioral: Health Belief Model (HBM) Based WhatsApp Oral Health Education Program — The program includes short educational videos, weekly thematic content, reminders, and behavior-reinforcement messages aimed at enhancing oral health knowledge, HBM constructs, and oral hygiene behaviors among individuals with Type 2 Diabetes Mellitus.
  Arms: Health Belief Model Based WhatsApp Oral Health Education Program
Behavioral: Educational Brochure Group — The Educational brochure provides information on the relationship between Type 2 Diabetes Mellitus and oral health and recommended oral hygiene practices. No WhatsApp based videos are provided during the study period
  Arms: Educational Brochure Group

SUMMARY:
The goal of this Educational interventional study is to test the usefulness of an educational program delivered through WhatsApp videos in increasing oral health knowledge and habits in people with Diabetes between the age of 18 and 65 years. The main question it aims to answer is:

Does a WhatsApp-based educational Program improve oral health knowledge and behaviors in people with diabetes, and is it more effective than education delivered through brochures? Participants in one group will receive educational videos through WhatsApp, while the other group receive a brochure containing oral health information. Researchers will then compare the groups to see if the intervention made a difference.

Participants will:

* Fill a baseline questionnaire to assess their current knowledge and behaviors.
* They then either participate in a one-month educational program delivered through WhatsApp, or receive an educational brochure.
* Wait for 1 month after the program to allow for application of knowledge.
* Fill a post intervention questionnaire to assess changes in knowledge and behavior.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether an educational intervention based on the Health Belief Model (HBM) and delivered through WhatsApp may improve diabetes patients' oral health behaviors and knowledge. This study is a randomized controlled trial (RCT) with two groups: an intervention group (WhatsApp-based education) and a control group (brochure-based education). Adults (18-65 years) with Type 2 Diabetes Mellitus from a diabetes clinic in Karachi were recruited. 98 participants (49 in each group) were selected through random allocation. The randomization process ensured that participants are evenly distributed between the groups based on key factors, specifically gender, educational level and duration of diabetes to reduce potential bias from these characteristics. This study was a single blinded study in which participants were not informed about the existence of two distinct groups. The WhatsApp based intervention consisted of 12 short educational videos, each approximately 3 to 5 minutes in duration, these videos were sent individually to each participant every alternate day from Monday to Friday, resulting in three videos per week over a period of one month, Reminders were sent the following day after each video to encourage engagement and sustain behavior change. Each week was focused on specific HBM constructs delivered through short, professionally scripted educational videos in Urdu. Each week was focused on specific HBM constructs. The control group received only an educational brochure.

A structured questionnaire was used to evaluate participants' knowledge and oral hygiene practices at two points: baseline (before intervention) and one-month post-intervention. The questionnaire was designed to measure HBM constructs (e.g. perceived susceptibility, severity, benefits, barriers, cues to action, and self-efficacy), awareness of oral care and oral hygiene related behaviors. Data were analyzed using SPSS Version 27.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years with a confirmed diagnosis of T2DM
* Able to use WhatsApp for the study duration
* Able to read and write in Urdu

Exclusion Criteria:

* Edentulous
* Individuals diagnosed with life-threatening diseases such as advanced cancer, end-stage renal disease, or severe cardiac failure
* Diminished cognitive ability
* Radiotherapy in head and neck region.
* Planning to migrate during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Oral Health Knowledge Score | Baseline and 4 weeks after intervention
  The participant's knowledge about the relationship between diabetes and oral health issues, will be assessed through a structured Questionnaire consisting of 10 binary items. (Yes = 1, No = 0). A total knowledge score ranging from 0 to 10 will be calculated by summing item responses, with higher scores indicating greater oral health knowledge. Pre- and post-knowledge scores will be compared, and cutoff scores will be calculated using the mean and Standard Deviation.

SECONDARY OUTCOMES:
Health Belief Model Construct Scores | Baseline and 4 weeks after intervention
  Health Belief Model constructs, including perceived susceptibility, perceived severity, perceived benefits, perceived barriers, self-efficacy, and cues to action, will be assessed using a structured Questionnaire. Items will be measured on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Separate construct scores will be calculated by summing item responses within each domain, with higher scores indicating stronger beliefs or perceptions related to oral health behaviors.
Oral Hygiene Behavior Score | Baseline and 4 weeks after intervention
  Participants' reported frequency and quality of oral health practices, including brushing, flossing, gingival health, and dental visits will be measured on a scale of 0(never) to 4(always) using a structured questionnaire. Higher scores indicate better oral hygiene-related behaviors. Pre- and post-intervention scores will be compared, and cutoff levels will be determined using the mean and standard deviation(SD).

CONTACTS AND LOCATIONS:
Overall Officials: ILMA KIRAN, BDS, MPH, Principal Investigator — Dow University of Health Sciences
Locations (1):
- National Institute of Diabetes & Endocrinology, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The study does not include a plan to make individual participant data (IPD) available due to privacy considerations and absence of participant consent for public data sharing.

REFERENCES:
- [Background] Jacome-Hortua AM, Rincon-Rueda ZR, Sanchez-Ramirez DC, Angarita-Fonseca A. Effects of a WhatsApp-Assisted Health Educational Intervention for Cardiac Rehabilitation: A Randomized Controlled Clinical Trial Protocol. Methods Protoc. 2024 Apr 19;7(2):35. doi: 10.3390/mps7020035. PMID 38668142
- [Background] Gao X, Wong ML, Kalhan AC, Xie JJ, Siti Hajar H, Yeo ABK, Allen PF. Theory-derived intervention to improve oral health of older adults: study protocol for a randomised controlled trial. BMJ Open. 2022 Dec 12;12(12):e064791. doi: 10.1136/bmjopen-2022-064791. PMID 36523250
- [Result] Jeihooni AK, Jamshidi H, Kashfi SM, Avand A, Khiyali Z. The Effect of Health Education Program Based on Health Belief Model on Oral Health Behaviors in Pregnant Women of Fasa City, Fars Province, South of Iran. J Int Soc Prev Community Dent. 2017 Nov-Dec;7(6):336-343. doi: 10.4103/jispcd.JISPCD_339_17. Epub 2017 Dec 29. PMID 29387617
- [Result] Omar MA, Hasan S, Palaian S, Mahameed S. The impact of a self-management educational program coordinated through WhatsApp on diabetes control. Pharm Pract (Granada). 2020 Apr-Jun;18(2):1841. doi: 10.18549/PharmPract.2020.2.1841. Epub 2020 May 3. PMID 32477434
- [Result] Haghdoost A, Bakhshandeh S, Tohidi S, Ghorbani Z, Namdari M. Improvement of oral health knowledge and behavior of diabetic patients: an interventional study using the social media. BMC Oral Health. 2023 Jun 3;23(1):359. doi: 10.1186/s12903-023-03007-w. PMID 37270487
- [Result] Malekmahmoodi M, Shamsi M, Roozbahani N, Moradzadeh R. A randomized controlled trial of an educational intervention to promote oral and dental health of patients with type 2 diabetes mellitus. BMC Public Health. 2020 Mar 4;20(1):287. doi: 10.1186/s12889-020-8395-4. PMID 32131790
- See also: Provides general information on the relationship between diabetes and oral health and guidance on maintaining good oral hygiene habits to prevent gum disease and oral complications. — https://diabetes.org/health-wellness/keeping-your-mouth-healthy
- See also: Provides concise information on how diabetes increases the risk of oral diseases such as gum infection and tooth decay, and emphasizes the importance of good oral hygiene and regular dental care as part of diabetes management. — https://idf.org/about-diabetes/diabetes-complications/diabetes-and-oral-health/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT07323771/Prot_SAP_000.pdf